CLINICAL TRIAL: NCT03004378
Title: The Role of Activity Tracking on Weight Loss in Obese Adolescents
Brief Title: Interventions for Adolescent Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0241
Record Dates: First submitted 2016-12-20; First posted 2016-12-28 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2018-04

CONDITIONS: Adolescent Obesity
Keywords: obesity; adolescent; tracking device; fitbit
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive the clinic standard of care which includes individual assessment and management by: a pediatric gastroenterologist, a pediatric surgeon, a dietitian, and a fitness instructor who are present at every visit.
- Intervention (Experimental): Fitbit (activity tracker) + participants will receive the clinic standard of care which includes individual assessment and management by: a pediatric gastroenterologist, a pediatric surgeon, a dietitian, and a fitness instructor who are present at every visit.
  Interventions: Behavioral: Activity Tracker

INTERVENTIONS:
Behavioral: Activity Tracker — Fitbit Alta
  Arms: Intervention

SUMMARY:
This study will evaluate whether the short-term use of activity tracking devices improves short-term weight loss in adolescents. The investigators will evaluate whether weight loss translates into a change in obesity-related biomarkers associated with adolescent obesity. In addition, the investigators will report outcomes after the implementation of activity tracking devices in conjunction with an intense adolescent weight loss program.

DETAILED DESCRIPTION:
This study will evaluate the short-term use of activity tracking devices and their effects on short- and long-term weight loss in adolescents. The investigators plan to establish whether weight loss translates into a change in obesity-related biomarkers associated with adolescent obesity. Each participant with an activity tracking device will have the goal of reaching 10,000 steps per day, in addition to their individual fitness plan.

ELIGIBILITY:
Inclusion Criteria:

Ages 12-18 years BMI ≥ 95th percentile for age and sex group Participant able to read and understand English Willingness to be randomized to any condition

Exclusion Criteria:

Inability to obtain informed parental consent and/or child assent Inability to participate in the program due to pre-existing conditions (e.g., paralysis, heart failure, severe autism or mental retardation, psychosis) Pregnancy Clinical judgment concerning safety Inability of the participant to speak English

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the pilot trial will be measured by an attrition rate of ≤50%. | 18 weeks
  We set a study attrition rate of participants at ≤50% as the feasibility measure for the study.

SECONDARY OUTCOMES:
Body mass index (BMI) (kg/m2) | Change from 0 to 18 weeks
  Absolute change in BMI
Weight (kg) | Change from 0 to 18 weeks
  Weight change
Change in obesity related biomarkers | Change from 0 to 18 weeks
  AST: aspartate aminotransferase; ALT: alanine aminotransferase; GGT: gamma glutamyl transferase; CRP: C reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Kanika K Bowen-Jallow, MD, MMS, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide all data, regardless of publication, collected as part of this project. All external investigators must submit a written request identifying their research question(s) and specifying the data they are requesting. The request must include a data security plan and explanation of how the data will be stored and who will have access.
Supporting Information: Study Protocol, SAP
Time Frame: Data will only be available upon request
Access Criteria: The request must include a data security plan and explanation of how the data will be stored and who will have access.

REFERENCES:
- [Derived] Bowen-Jallow K, Nunez-Lopez O, Wright A, Fuchs E, Ahn M, Lyons E, Jupiter D, Berry L, Suman O, Radhakrishnan RS, Glaser AM, Thompson DI. Wearable Activity Tracking Device Use in an Adolescent Weight Management Clinic: A Randomized Controlled Pilot Trial. J Obes. 2021 Jan 7;2021:7625034. doi: 10.1155/2021/7625034. eCollection 2021. PMID 33505717